CLINICAL TRIAL: NCT02487017
Title: Phase 2 Study of DC-CIK Cells Combined With TACE in the Treatment of Hepatocellular Carcinoma
Brief Title: DC-CIK Combined With TACE in the Treatment of Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Hornetcorn Bio-technology Company, LTD (Industry)
Collaborators: Yantai City Hospital for Infectious Diseases (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYK-Hepatocellular Carcinoma
Record Dates: First submitted 2015-06-29; First posted 2015-07-01 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2015-12

CONDITIONS: Hepatocellular Carcinoma; Neoplasms; Digestive System Neoplasms
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasms; Digestive System Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transcatheter Arterial Chemoembolization (Sham Comparator): Transcatheter Arterial Chemoembolization treatment according to NCCN guidelines，patients will receive 5-FU Hepatic arterial infusion,3 cycles at least.
  Interventions: Procedure: Transcatheter Arterial Chemoembolization (TACE)
- DC-CIK (Experimental): After accepting concurrent TACE according to NCCN guidelines,patients will receive 3 cycles of DC-CIK treatment at least.
  Interventions: Biological: DC-CIK

INTERVENTIONS:
Procedure: Transcatheter Arterial Chemoembolization (TACE) — Transcatheter Arterial Chemoembolization (TACE):
  5-FU 400mg/m2 Hepatic arterial infusion ,lipiodol amount is usually 20 ml,the perfusion time should not be less than 20 min
  Arms: Transcatheter Arterial Chemoembolization
Biological: DC-CIK — Transcatheter Arterial Chemoembolization (TACE):
  5-FU 400mg/m2 Hepatic arterial infusion ,lipiodol amount is usually 20 ml, the perfusion time should not be less than 20 min
  DC-CIK:
  8×10^9 DC-CIK cells for each infusion, IV (in the vein) for each infusion at least 3 cycles, each cycle received four infusions on day 14, 16, 30 and 32
  Arms: DC-CIK

SUMMARY:
Evaluation of DC-CIK cells combined TACE treatment for HCC

DETAILED DESCRIPTION:
60 patients with Hepatocellular Carcinoma, who had received Transcatheter Arterial Chemoembolization (TACE) , will be randomly divided into group A (receive DC-CIK+ TACE treatment) or group B (just receive TACE), and the randomize ratio will be 1:1.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old;
* Histologically confirmed with Hepatocellular Carcinoma at stage I-II;
* Patients who can accept Transcatheter Arterial Chemoembolization ;
* Patients who have a life expectancy of at least 3 months;
* Patients who have a Child-Pugh:A/B; .Eastern Cooperative Oncology Group (ECOG) performance status was 0-2.

Exclusion Criteria:

* White blood cell <3 x 10^9/L,Platelet count <75 x 10^9/L;BUN and Cr more than normal limits on 3.0 times ;
* Known or suspected allergy to the investigational agent or any agent given in association with this trial;
* Pregnant or lactating patients;
* Known history of Human Immunodeficiency Virus (HIV), Hepatitis C Virus (HCV) or TreponemaPallidun (TP) infection;
* Patients who are suffering from serious autoimmune disease;
* Patients who had used long time or are using immunosuppressant;
* Patients who had active infection;
* Prior use of any anti-cancer treatment in 30 days;
* Now or recently will join another experimental clinical study ;
* History of organ allograft;
* Other situations that the researchers considered unsuitable for this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3 years

SECONDARY OUTCOMES:
Progress-free survival | 3 years
Quality of life (QOL) | 3 years
Phenotypic analysis of T cells | 1 years

CONTACTS AND LOCATIONS:
Overall Officials: Xiangzhong Liu, Professor, Principal Investigator — Yantai City Hospital for Infectious Diseases Immunotherapy center
Locations (1):
- Yantai City Hospital for Infectious Diseases, Yantai, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided